CLINICAL TRIAL: NCT02423902
Title: A Single-arm, Open-label Study of Ad-RTS-hIL-12 + Veledimex Following First-, Second-, or Third-Line Standard Treatment in Subjects With Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Ad-RTS-hIL-12 With Veledimex in Subjects With Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated after 9 subjects had enrolled under Protocol Amend 1 because of slower than expected accrual. Protocol Amendment 2 (16 May 2016) was submitted to the FDA and, based on the decision of the PI, was not submitted to the IRB.
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI001-203
Record Dates: First submitted 2015-04-06; First posted 2015-04-22 (Estimated); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — veledimex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ad-RTS-hIL-12 + Veledimex (Experimental): Intratumoral injection of Ad-RTS-hIL-12 in combination with veledimex
  Interventions: Biological: Ad-RTS-hIL-12; Drug: Veledimex

INTERVENTIONS:
Biological: Ad-RTS-hIL-12 — Approximately 1.0x10^12 viral particles (vp) per injection
  Other Names: INXN-2001
Drug: Veledimex — 7 oral doses of veledimex
  Other Names: INXN-1001 (activator ligand)

SUMMARY:
This is a single-arm, phase Ib/II study to examine the safety, tolerability and preliminary efficacy of one cycle of Ad-RTS-hIL-12 immunotherapy in women with advanced breast cancer and pre-study SD or PR after completion of a minimum 12 week course of standard first- or second-line chemotherapy. The patient population will include patients with locally advanced or metastatic breast cancer of all subtypes.

DETAILED DESCRIPTION:
Subjects who have PD or a CR after the standard chemotherapy are not eligible for the study. Following entry into the trial, patients will go on a treatment holiday from chemotherapy and enter an immunotherapy phase of treatment. Continuation of HER2-targeted antibody therapy is permitted during this immunotherapy phase for women with HER2+ disease. Scans will be conducted at 6 and 12 weeks after the start of Ad-RTS-hIL-12 immunotherapy to determine tumor response. Radiographic PD at week 6 must be confirmed at least 4 weeks later, either at week 12 or earlier if clinically necessitated.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥ 18 years
2. Histologically-confirmed, locally advanced or metastatic adenocarcinoma of the breast
3. Achievement of SD or PR after a minimum of 12 weeks of pre-study first- or second-line standard chemotherapy
4. Presence of at least 2 measurable lesions
5. Standard treatment interrupted, except if anti-HER2 therapy
6. All treatment-related or radiation-related toxicities resolved to Grade 1 or lower
7. Submission of copies of tumor measurements and scans
8. Life expectancy > 12 weeks
9. ECOG performance status of 0 to 1
10. Adequate bone marrow function
11. Adequate liver function
12. Adequate renal function
13. Female subjects and their male partners must agree must agree to use a highly reliable method of birth control
14. Able to swallow oral medication
15. Willing to comply with study procedures

Exclusion Criteria:

1. Metastatic breast cancer patients currently on hormonal therapy as first- or second-line are not permitted
2. Prior radiation therapy encompassing > 25% of bone marrow
3. Any congenital or acquired condition leading to compromised ability to generate an immune response
4. Immunosuppressive therapy

   1. Use of systemic immunosuppressive drugs
   2. Requirement for continual immune suppression
5. Major surgery within 4 weeks of study treatment
6. An active, second potentially life-threatening cancer
7. Presence of brain or subdural metastases

   1. Any signs and/or symptoms of brain metastases must be stable for ≥ 4 weeks
   2. Radiographic stability should be determined by comparing contrast-enhanced CT or MRI scans at screening to scans obtained by the same method at least 4 weeks earlier
8. Presence or documented history of any of the following autoimmune conditions:

   1. Inflammatory bowel disease
   2. Rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis
   3. Motor neuropathy considered of autoimmune origin
9. Presence of meningeal carcinomatosis
10. Use of any medications that induce, inhibit, or are substrates of CYP450 3A4
11. History or evidence of cardiac disease as indicated by any of the following:

    1. Congestive heart failure greater than NYHA Class II
    2. Unstable angina or new-onset angina (begun within the last 3 months), or myocardial infarction within the 6 months prior to enrollment
    3. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
    4. Congenital long QT syndrome or taking drugs known to prolong the QT interval
12. Current use of any drugs with a known risk of causing torsades de pointes
13. Evidence or history of thromboembolic, venous, or arterial events within the past 3 months
14. Evidence or history of bleeding diathesis or coagulopathy
15. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) > 1.5 x ULN, in subject who is not therapeutically anticoagulated.
16. History of malabsorption syndrome or other condition that would interfere with enteral absorption
17. Presence of active clinically serious infection
18. Diagnosis of infection with HIV or chronic infection with hepatitis B or C
19. Any other unstable or clinically significant concurrent medical condition
20. Pregnant or breast-feeding
21. Use of any investigational, non-United States Food and Drug Administration (US FDA) approved drug
22. Participation in any other clinical trial
23. Presence of any condition which makes the patient unsuitable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07-18 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HER2+ Subjects: Subjects with HER2+ breast cancer were assigned to receive an intratumoral injection of Ad-RTS-hIL-12 in combination with veledimex:
  * Ad-RTS-hIL-12: Approximately 1.0x10^12 viral particles (vp) per injection
  * Veledimex: 7 oral doses of veledimex
- HER2- Subjects: Subjects with HER2- breast cancer were assigned to receive an intratumoral injection of Ad-RTS-hIL-12 in combination with veledimex:
  * Ad-RTS-hIL-12: Approximately 1.0x10^12 viral particles (vp) per injection
  * Veledimex: 7 oral doses of veledimex
Period: Overall Study
Arm/Group | HER2+ Subjects | HER2- Subjects
Started | 1 | 8
Completed | 0 | 4
Not Completed | 1 | 4
Not completed — Disease progression | 1 | 4

BASELINE CHARACTERISTICS:
Population: The safety population will comprise all subjects who have received either the injection of Ad-RTS-hIL-12 or any doses of veledimex
Groups:
- Total: Total of all reporting groups
Arm/Group | HER2+ Subjects | HER2- Subjects | Total
Number analyzed (Participants) | 1 | 8 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (0) | 50.9 (10.24) | 49.6 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 7 | 8
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 6 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 167.0 (0) | 161.1 (4.72) | 161.8 (4.83)
Weight [Mean (Standard Deviation); unit: kg] | 71.0 (0) | 63.2 (11.75) | 64.1 (11.29)
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.5 (0) | 24.5 (5.02) | 24.6 (4.71)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events Leading to Study Discontinuation
Description: Composite measure of safety and tolerability based on lab parameters, vitals, physical examination data and deaths, SAEs, and AEs resulting in patient discontinuation. Toxicity stopping rules when applicable will be determined based on a clinical assessment made by the SRC.
  The Sponsor conducted an additional ad hoc analysis of study-drug-related-TEAEs with an onset during the dosing period of all cycles to assess the number subjects with events of cytokine release syndrome (CRS), to include TEAEs that were symptoms of CRS, including when the PI did not report the preferred term of CRS. Results of this ad hoc assessment are reported here.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
participants
  Any TEAE | 1 | 8
  Treatment-related TEAE | 1 | 8
  Grade 3 or higher TEAE | 1 | 7
  Treatment-related Grade 3 or higher TEAE | 1 | 6
  Adverse event leading to death | 0 | 0
  Serious TEAE | 0 | 4
  TEAE leading to discontinuation | 0 | 5
  Cytokine Release Syndrome Assessment: Grade 2 | 1 | 5
  Cytokine Release Syndrome Assessment: Grade 3 | 0 | 2
  Cytokine Release Syndrome Assessment: Grade 4 | 0 | 1

2. Secondary Outcome: Progression Rate at 12 Weeks After the Start of One Cycle of Ad-RTS-hIL-12 Immunotherapy
Description: The percent of subjects that failed by 12 weeks is denoted as the progression rate, and is derived based on the sum of progression events, death events, and subjects who discontinue the trial due to an AE. Tumor assessment was performed per RECIST (progression was determined as >=20% increase in the sum of the longest diameter of target lesions and or unequivocal new lesion were present)
Time Frame: 12 weeks
Population: The veledimex-treated population will comprise subjects who have received the injection of Ad-RTS-hIL-12 and at least one dose of veledimex
Measure: Number (95% Confidence Interval); unit: % of subjects who progressed at 12 weeks
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
% of subjects who progressed at 12 weeks
  12-week Progression rate per RECIST criteria | 100.0 [2.5 to 100.0] | 62.5 [24.5 to 91.5]
  12-week Progression rate per irRC criteria | 100.0 [2.5 to 100.0] | 75.0 [34.9 to 96.8]

3. Secondary Outcome: Overall Response Rate (ORR), Defined as the Rate of Complete Response (CR) Plus the Rate of Partial Response (PR) at 12 Weeks Following the Start of Ad-RTS-hIL-12 Immunotherapy
Description: Overall response at Week 12 is based on the totality of the responses for target and non-target lesions. For this calculation, responders are defined as those experiencing a CR or a PR. Non-responders are those either with stable or progressive disease. Those subjects who cannot be assessed will be treated as non-responders for the purposes of deriving the percentage of responders and confidence intervals.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects with CR or PR
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
Percentage of subjects with CR or PR
  Objective response rate (CR or PR) at Week 12 per RECIST | 0.0 [0.0 to 97.5] | 12.5 [0.3 to 52.7]
  Objective response rate (CR or PR) at Week 12 per irRC | 0.0 [0.0 to 97.5] | 12.5 [0.3 to 52.7]

4. Secondary Outcome: Disease Control Rate (DCR), Defined as the Proportion of Subjects Who Have a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) at 12 Weeks Following the Start of One Cycle of Ad-RTS-hIL-12 Immunotherapy
Description: The DCR is the proportion of subjects who have a CR, PR, or stable disease at 12 weeks following the start of Ad-RTS-hIL-12 immunotherapy using RECIST v1.1. For this calculation, responders are defined as those experiencing a CR, PR, or stable disease. Non-responders are defined as those with PD. Those subjects that cannot be assessed will be treated as non-responders for the purposes of deriving the percentage of responders and confidence intervals.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects with CR, PR, or S
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
Percentage of subjects with CR, PR, or S
  Disease control rate (CR, PR, or SD) at Week 12 per RECIST | 0.0 [0.0 to 97.5] | 25.0 [3.2 to 65.1]
  Disease control rate (CR, PR, or SD) at Week 12 per irRC | 0.0 [0.0 to 97.5] | 25.0 [3.2 to 65.1]

5. Secondary Outcome: Number of Subjects Whose Baseline Tumor Status (Stable Disease or Partial Response) Improves to Partial Response or Better at 12 Weeks Following the Start of Ad-RTS-hIL-12 Immunotherapy
Description: Number of subjects whose baseline tumor status (stable disease or partial response) improves to partial response or better at 12 weeks following the start of Ad-RTS-hIL-12 immunotherapy
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
participants | 0 | 1

6. Secondary Outcome: Comparison of Radiographic Tumor Responses by irRC With RECIST
Description: Best Overall Response at Week 12 after 1 cycle of Ad-RTS-hIL-12 + veledimex immunotherapy is reported for response assessment per RECIST and per irRC.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
participants
  Partial response per RECIST | 0 | 1
  Partial response per irRC | 0 | 1
  Stable disease per RECIST | 0 | 3
  Stable disease per irRC | 0 | 2
  Progressive disease per RECIST | 1 | 4
  irRProgressive disease per irRC | 1 | 5

7. Secondary Outcome: Change From Baseline in Serum CA15-3 Levels
Description: Serum levels of the cancer antigen 15-3 (CA15-3) biomarker were measured by immunoassay to explore the impact of treatment.
Time Frame: Screening, Week 6, and Week 12
Population: The analysis was performed on the Veledimex-treated population. The number of subjects analyzed at each time point may be lower than the total due to missed sample collections.
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
U/ml
  CA15-3 (Muc-1) at Screening | 91 (0) | 1281.5 (3500.774)
  CA15-3 (Muc-1) at Week 6 | 138 (0) | 3747.5 (10430.77)
  CA15-3 (Muc-1) at Week 12: number analyzed (Participants) | 0 | 4
  CA15-3 (Muc-1) at Week 12 |  | 76.75 (101.6772)

8. Secondary Outcome: Change From Baseline in Serum Interleukin-12 (IL-12) Levels
Description: Serum levels of Interleukin-12 (IL-12) were measured by immunoassay to explore the impact of treatment on immune biomarkers.
Time Frame: Screening, Week 6, and Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
pg/mL
  Il-12 at Screening | 0.1505 | 0.0728 (0.0901)
  Il-12 at Week 6: number analyzed (Participants) | 1 | 7
  Il-12 at Week 6 | 0.735 | 0.1476 (0.1436)
  Il-12 at Week 12: number analyzed (Participants) | 0 | 4
  Il-12 at Week 12 |  | 0.0244 (0.0221)

9. Secondary Outcome: Change From Baseline in Serum Interferon-gamma (IFN-gamma) Levels
Description: Serum levels of Interferon-gamma (IFN-gamma) were measured by immunoassay to explore the impact of treatment on immune biomarkers.
Time Frame: Screening, Week 6, and Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
pg/mL
  IFN-gamma at Screening | 6.34 | 7.34 (10.32)
  IFN-gamma at Week 6 | 6.87 | 6.51 (6.06)
  IFN-gamma at Week 12: number analyzed (Participants) | 0 | 4
  IFN-gamma at Week 12 |  | 7.02 (6.24)

10. Secondary Outcome: Change From Baseline in Serum Carcinoembryonic Antigen (CEA) Levels
Description: Serum levels of the carcinoembryonic antigen (CEA) biomarker were measured by immunoassay to explore the impact of treatment.
Time Frame: Screening, Week 6, and Week 12.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HER2+ Subjects | HER2- Subjects
Number analyzed (Participants) | 1 | 8
ng/mL
  CEA at Screening | 5.1 | 8.275 (9.970)
  CEA at Week 6 | 7.5 | 14.838 (21.690)
  CEA at Week 12: number analyzed (Participants) | 0 | 4
  CEA at Week 12 |  | 4.225 (3.226)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HER2+ Subjects | HER2- Subjects
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/1 | 4/8
Other Adverse Events (participants affected / at risk) | 1/1 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER2+ Subjects (N=1) | HER2- Subjects (N=8)
Febrile Neutropenia (Blood and lymphatic system disorders) | NA | 1 (1)
Fatigue (General disorders) | NA | 2 (2)
Malaise (General disorders) | NA | 2 (2)
Lung Infection (Infections and infestations) | NA | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | NA | 1 (1)
Alanine Aminotransferase Increased (Investigations) | NA | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | NA | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Hypotension (Vascular disorders) | NA | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER2+ Subjects (N=1) | HER2- Subjects (N=8)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 6 (9)
Fatigue (General disorders) | 1 (1) | 5 (8)
Chills (General disorders) | 1 (1) | 5 (6)
Malaise (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Localised Oedema (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (2) | 2 (2)
Alanine Aminotransferase (Investigations) | 1 (1) | 2 (2)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 4 (4)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 2 (2)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT02423902/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT02423902/SAP_001.pdf